CLINICAL TRIAL: NCT00702195
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established During Phase II Clinical Trials for the Development of Org 36286 (Corifollitropin Alfa).
Brief Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established During Phase II Clinical Trials of Org 36286 (Study 38817)(P06054)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P06054; 38817
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy
Keywords: Neonatal outcome; Congenital malformations; In-Vitro Fertilization; Controlled ovarian stimulation; Follow-up; Ovulation Induction; Neonates
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Experimental Group 1: all doses of Org 36286 (corifollitropin alfa) from trial 38805 (7.5 μg, 15 μg, 30 μg and 60 μg)
  Interventions: Drug: Org 36286 (corifollitropin alfa)
- Experimental Group 2: Placebo
  Interventions: Drug: Placebo
- Experimental Group 3: all doses of Org 36286 (corifollitropin alfa) from trial 38807 (120 μg, 180 μg and 240 μg)
  Interventions: Drug: Org 36286 (corifollitropin alfa)
- Experimental Group 4: 150 IU Puregon®
  Interventions: Drug: recFSH

INTERVENTIONS:
Drug: Org 36286 (corifollitropin alfa) — single dose of Org 36286 (corifollitropin alfa) administered under protocol 38805/38807
  Other Names: corifollitropin alfa
  Groups: Experimental Group 1; Experimental Group 3
Drug: Placebo — single dose of placebo (administered under protocol 38805)
  Groups: Experimental Group 2
Drug: recFSH — 150 IU recFSH daily (reference group administered under protocol 38807)
  Other Names: follitropin beta; Puregon®; Follistim®
  Groups: Experimental Group 4

SUMMARY:
The objective of this trial was to evaluate whether Org 36286 treatment in any Phase IIa clinical development trial of Org 36286 for OI or COH in assisted reproductive treatment programs was safe for pregnant subjects and their offspring. Data from subjects who participated in Trials 38805 and 38807 and became pregnant were evaluated.

DETAILED DESCRIPTION:
This was an open prospective follow-up trial to monitor pregnancy, delivery, and neonatal outcome of women who became pregnant during any Phase IIa clinical trial of Org 36286 for OI or COH for IVF. For this trial, no study specific assessments were required, but information obtained in standard practice was used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects taking part in any clinical development trial of Org 36286 for OI or COH for IVF in Phase IIa;
* Ongoing pregnancy confirmed by ultrasonography (USS) at or beyond 12 weeks of gestation;
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women who became pregnant during Trials 38805 or 38807 were enrolled in Trial 38817
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2003-09-15 (Actual); Study Completion 2003-09-15 (Actual)

PRIMARY OUTCOMES:
Pregnancy status at 20 weeks of gestation; Take-home baby rate | one pregnancy period

SECONDARY OUTCOMES:
Pregnancy follow-up; Delivery follow-up; Neonatal outcome; Infant follow-up; Congenital Malformations and Chromosomal Abnormalities | one pregnancy period

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997